CLINICAL TRIAL: NCT05675475
Title: Study of the Association Between Digital Eye Syndrome With Binocular Vision and the Ocular Surface in Higher Education Students in the Area of Health Technologies
Acronym: DESIROUS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universidade Nova de Lisboa (Other)
Collaborators: NOVA Medical School | Faculdade de Ciências Médicas, Universidade Nova de Lisboa (Unknown); Escola Superior de Tecnologia da Saúde de Lisboa (ESTeSL) (Unknown); University of Évora (Other); CINTESIS@RISE, NOVA Medical School | Faculdade de Ciências Médicas, Universidade Nova de Lisboa (Unknown); Comprehensive Health Research Center (CHRC), Universidade Nova de Lisboa (Unknown)
Responsible Party: Sponsor
Other Study IDs: DESIROUS
Record Dates: First submitted 2022-12-12; First posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-12

CONDITIONS: Digital Eye Strain
Keywords: accommodation; convergence; tear film

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Exposure — Higher education students from health technologies field exposed to digital devices.
Diagnostic Test: Orthoptic assessment (Outcome measure) — The orthoptic assessment is a non-invasive assessment that will last for 30 min to determine visual parameters related to binocular vision. It will be carried out by the research team in the orthoptics and vision sciences laboratories of the Lisbon School of Health Tecnology.
Diagnostic Test: Tear film Break Up Time (BUT) test (Outcome measure) — The BUT test is a tear film rupture assessment test that allows the stability of the tear film to be evaluated. To perform these tests, it is necessary to instill fluorescein and then it is observed in the slit lamp under illumination with a cobalt blue filter, to count the break-up time.

SUMMARY:
The goal of this observational study is to determinate the association between DES and changes in binocular vision and ocular surface. in higher education students in the area of health technologies. The main questions it aims to determine the prevalence of Digital Eye Syndrome (DES); the association between DES and changes in binocular vision and ocular surface; whether the time of use and the type of electronic devices influences the degree and type of symptoms of DES; and to determine whether there is an association between the type of ametropia and the symptoms of DES. Participants will have to answer 3 questionnaires (the Computer Vision Syndrome Questionnaire; the Convergence Insufficiency Symptoms Survey, and the Dry Eye Questionnaire (DEQ-5)) and then they will perform an orthoptic assessment and an assessment of the ocular surface with the tear film Break Up Time (BUT) test.

ELIGIBILITY:
Inclusion Criteria:

* Students of the first, second and third year of the degrees offered by Lisbon School of Health Technology, Instituto Politécnico de Lisboa;
* Age between 18 to 39 years;
* Accept and sign the consent.

Exclusion Criteria:

* Working Students;
* Students with known binocular vision disorders;
* Previous eye surgeries.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Higher Education Students in the Area of Health Technologies.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Digital Eye Syndrome | Immediately after subject enrollment, up to 1 week (single point collection)
  To verify the existence or absence of digital fatigue syndrome in higher education students. For this purpose, the Computer Vision Syndrome Questionnaire will be used. To verify the existence or not of digital fatigue syndrome in higher education. The Computer Vision Syndrome Questionnaire (CVS-Q) will be applied, which is composed of 16 x 2 questions, to assess the symptoms and their intensity. This questionnaire makes it possible to classifying CVS as asymptomatic and symptomatic.

SECONDARY OUTCOMES:
Convergence Insufficiency Symptoms Survey | Immediately after subject enrollment, up to 1 week (single point collection)
  The main objective of this questionnaire is to assess the frequency of symptoms of visual discomfort and consists of fifteen questions. The answers to the questions are evaluated and allow classifying binocular vision into "norm", "suspected convergence insufficiency" and "convergence insufficiency".
Dry Eye Questionnaire (DEQ-5) | Immediately after subject enrollment, up to 1 week (single point collection)
  The DEQ-5 questionnaire is the reduced version of the DEQ questionnaire that allows the assessment of dry eye. this questionnaire is made up of 5 questions and allows to obtain an answer score that classifies as "normal" and "dry eye".
Far Visual Acuity | Immediately after subject enrollment, up to 1 week (single point collection)
  Visual acuity is the spatial resolution capability of the visual system. The unit of measurement for this variable will be the minimum resolution angle algorithm (LogMAR).
Near Visual Acuity | Immediately after subject enrollment, up to 1 week (single point collection)
  Visual acuity is the spatial resolution capability of the visual system. The unit of measurement for this variable will be the minimum resolution angle algorithm (LogMAR).
Far Cover Test | Immediately after subject enrollment, up to 1 week (single point collection)
  The cover test is one of the variables used to study the motor component of the visual system and is a categorical variable, which will allow the identification of latent and manifest ocular deviations.
Near Cover Test | Immediately after subject enrollment, up to 1 week (single point collection)
  The cover test is one of the variables used to study the motor component of the visual system and is a categorical variable, which will allow the identification of latent and manifest ocular deviations.
Near Stereopsis | Immediately after subject enrollment, up to 1 week (single point collection)
  Stereopsis is one of the binocular vision parameters and the measurement unit used will be the arc seconds.
Near Point of Convergence | Immediately after subject enrollment, up to 1 week (single point collection)
  The near point of convergence is one of the convergence assessment methods and the unit of measurement is cm.
Flexibility of Accommodation | Immediately after subject enrollment, up to 1 week (single point collection)
  The flexibility of accommodation is one of the accommodation evaluation parameters and its measurement unit is cycle per minute.
Amplitude of Accommodation | Immediately after subject enrollment, up to 1 week (single point collection)
  The amplitude of accomodation is one of the accommodation evaluation parameters and its measurement unit is diopters.
Far Convergence | Immediately after subject enrollment, up to 1 week (single point collection)
  The far convergence is one of the elements of fusional vergencies and its measurement unit is the prismatic diopters.
Near Convergence | Immediately after subject enrollment, up to 1 week (single point collection)
  The near convergence is one of the elements of fusional vergencies and its measurement unit is the prismatic diopters.
Near Divergence | Immediately after subject enrollment, up to 1 week (single point collection)
  The near divergence is one of the elements of fusional vergencies and its measurement unit is the prismatic diopters.
Far Divergence | Immediately after subject enrollment, up to 1 week (single point collection)
  The far divergence is one of the elements of fusional vergencies and its measurement unit is the prismatic diopters.
Break Up Time Test | Immediately after subject enrollment, up to 1 week (single point collection)
  The BUT Test will allow assessing the stability of the tear film and the unit of measurement will be seconds.
Refrative Error | Immediately after subject enrollment, up to 1 week (single point collection)
  The refractive error will be assessed using the auto refratometer and your measurements will be in diopters.

CONTACTS AND LOCATIONS:
Overall Officials: André Rosário, PhD, Principal Investigator — NOVA Medical School | Faculdade de Ciências Médicas, Universidade Nova de Lisboa; Carla Lança, PhD, Principal Investigator — Escola Superior de Tecnologia da Saúde de Lisboa (ESTeSL)
Locations (1):
- Escola Superior de Tecnologia de Saúde de Lisboa, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No